CLINICAL TRIAL: NCT07059637
Title: Implementation of a Sarcopenia Clinic to Diagnose and Treat Skeletal Muscle Loss Due to COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Amy Attaway, Assistant Professor of Medicine, The Cleveland Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-857
Record Dates: First submitted 2025-07-08; First posted 2025-07-11 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: COPD; Emphysema; Sarcopenia
Keywords: COPD; emphysema; sarcopenia
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sarcopenia clinic (Active Comparator): Multidisciplinary sarcopenia clinic
  Interventions: Other: Multidisciplinary clinic evaluation
- COPD standard of care clinic (Active Comparator)
  Interventions: Other: COPD standard of care

INTERVENTIONS:
Other: Multidisciplinary clinic evaluation — The goal is to use evidence-based strategies to diagnose and treat sarcopenia due to COPD. The investigators anticipate that the approach will improve clinical outcomes for COPD patients with sarcopenia as compared to standard of care visits in ambulatory COPD clinics. The investigators will determine if the approach improves skeletal muscle mass and function, and also improves clinical outcomes related to frequency of hospitalizations, COPD exacerbations, or mortality. The approach is different than standard of care COPD treatment because it is informed by quantifying muscle mass and strength (through handgrip strength and bio-impedance) and have strong collaborations with nutrition and pulmonary rehabilitation.
  Arms: Sarcopenia clinic
Other: COPD standard of care — Standard COPD care treatment in an ambulatory post-hospital follow up clinic
  Arms: COPD standard of care clinic

SUMMARY:
Sarcopenia, or skeletal muscle loss, impacts up to 40% of COPD patients and is a major cause for morbidity and mortality. Despite the high clinical significance of sarcopenia in COPD, the diagnosis remains elusive because accurate measures of skeletal muscle are not tested during routine clinical care. The goal is to use evidence-based strategies to diagnose and treat sarcopenia due to COPD. The multidisciplinary team includes a pulmonologist, pharmacist, COPD nurse, and COPD coordinator. The investigators anticipate that the approach will improve clinical outcomes for COPD patients with sarcopenia as compared to standard of care visits in ambulatory COPD clinics. The investigators will determine if the approach improves skeletal muscle mass and function, and also improves clinical outcomes related to frequency of hospitalization or ED (Emergency Department) visits, COPD exacerbations, and mortality.

DETAILED DESCRIPTION:
The goal of this study is to determine whether the multidisciplinary sarcopenia clinic improves outcomes compared to standard of care ambulatory COPD clinics. The proposed study will be a prospective observational study. The investigators will compare the sarcopenia clinic with COPD ambulatory clinics and match based on severity of COPD. With informed consent and approval from Cleveland Clinic's IRB, the investigators will enroll patients with spirometry-confirmed COPD and evidence of sarcopenia who were recently admitted to either main campus Cleveland Clinic or regional facilities for a COPD exacerbation. COPD patients will be seen as a hospital follow up appointment in the multidisciplinary sarcopenia clinic or an outpatient ambulatory COPD clinic. Patients will be followed longitudinally for one year.

Subject Selection:

Recruitment: COPD patients admitted for a COPD exacerbation will be enrolled. Patients who are eligible for the trial will be offered placement in either the multidisciplinary clinic or the standard ambulatory COPD clinics. Our statistical analysis plan will include adjustment for disease severity using regression models, so that the same acuity of disease is being studied across both clinics.

ELIGIBILITY:
Inclusion Criteria:

1. COPD exacerbation as the primary cause for inpatient hospitalization OR secondary diagnosis of COPD exacerbation with acute respiratory failure as the primary diagnosis.
2. Patients must have CT (Computed Tomography) imaging performed during their admission and evidence of low skeletal muscle mass determined by CT imaging of the pectoralis muscle
3. Age > 40 years old.
4. Spirometry diagnosed COPD with FEV1/FVC ratio <0.70 with at least moderate obstruction (FEV1; forced expiratory volume in 1 second <80%).
5. Patients must have smoked at least 10 pack years and may be current or former smokers.

Exclusion Criteria:

1. History of other comorbid lung disease (i.e. interstitial lung disease, asthma).
2. Currently being evaluated or already listed for lung transplant.
3. Active malignancy.
4. Significant comorbid end organ failure defined as congestive heart failure (ejection fraction<40%), end stage renal disease requiring dialysis, or cirrhosis (based on radiologic imaging).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | One year follow up
  Count
Hospitalizations | One year follow up
  Count
Number of COPD exacerbations | One year follow up
  Count

SECONDARY OUTCOMES:
Handgrip strength | One year follow up
  kg
Skeletal muscle mass by bioelectric impedance analysis | One year follow up
  kg/m^2
6-minute walk distance | One year follow up
  meters

CONTACTS AND LOCATIONS:
Overall Officials: Amy Attaway, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
The data cannot be sufficiently de-identified to protect participant confidentiality due to small sample size.